CLINICAL TRIAL: NCT01906359
Title: The Acute Effects of Triacylglycerol Structure of Dietary Fats on Gut Hormones and Haemostatic Markers in Subjects With Type 2 Diabetes Mellitus
Brief Title: Effects of Triacylglycerol Structure on Gut Hormones and Haemostatic Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: Universiti Putra Malaysia (Other); Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: A005/11; NMRR-12-146-11363 (Registry Identifier: National Medical Research Register)
Record Dates: First submitted 2013-07-11; First posted 2013-07-24 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Interesterified fat; Stereospecific number 2; Gut hormones; GIP; Insulin sensitivity; Postprandial lipaemia; Haemostatic markers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dietary fat - PO (Experimental): Native palm olein (IV56)
  Interventions: Other: Native palm olein (IV56)
- Dietary fat - IPO (Experimental): Chemically interesterified palm olein (IV56)
  Interventions: Other: Chemically interesterified palm olein (IV56)
- Dietary fat - HOS (Experimental): High oleic sunflower oil
  Interventions: Other: High oleic sunflower oil

INTERVENTIONS:
Other: Native palm olein (IV56) — Test meal consists of a high fat muffin (containing 50 g native palm olein) and a cup of milkshake, to be taken as breakfast for each postprandial study day.
  Other Names: PO
  Arms: Dietary fat - PO
Other: Chemically interesterified palm olein (IV56) — Test meal consists of a high fat muffin (containing 50 g chemically interesterified palm olein) and a cup of milkshake, to be taken as breakfast for each postprandial study day.
  Other Names: IPO
  Arms: Dietary fat - IPO
Other: High oleic sunflower oil — Test meal consists of a high fat muffin (containing 50 g high oleic sunflower oil) and a cup of milkshake, to be taken as breakfast for each postprandial study day.
  Other Names: HOS
  Arms: Dietary fat - HOS

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a chronic disorder determined by lifestyle and genes. It is associated with chronic hyperglycaemia along with other metabolic abnormalities. It is also one of the risk factors for cardiovascular disease (CVD). This disease is due to insulin resistance and/or deficiency as well as increased hepatic glucose output. According to the Third National Health and Morbidity Survey (3rd NHMS), the prevalence of T2DM for adults aged 30 years and above is 14.9%, increased by almost 80% from 1996 to 2006. Dietary composition may affect insulin sensitivity, postprandial triacylglycerol concentration and the risk of T2DM. The role of dietary fats in T2DM is of particular interest and has been clinically studied for many decades. The type of fat we ingest every day consists of different types of fatty acids and different degree of saturation, which in turn influence glucose metabolism by altering cell membrane function, enzyme activity, insulin signalling and gene expression. Previous studies demonstrated that interesterification of dietary fat alter postprandial lipaemia. Saturated fat such as palm olein has been reported to display lower postprandial lipaemia after interesterification. Changing the structure of triacylglycerol (TAG) alters the physical properties of dietary fat which affects digestibility, metabolism and atherogenicity. A recent study conducted by Sanders and co-workers demonstrated reduced levels of plasma glucose-dependent insulinotropic polypeptide (GIP) following both the lard and interesterified palm olein (IPO) compared with the palm olein (PO) and high oleic sunflower oil (HOS) diets in healthy subjects. The GIP and glucagon-like peptide-1 (GLP-1) are major players in the modulation of postprandial insulin secretion by the pancreas. Although GIP secretion in response to meals is normal in patients with Type 2 diabetes mellitus (T2DM), GIP induced secretion of insulin is defective in diabetes. This is observed to be predominantly a defective stimulation of the late phase of insulin response (20-120 minutes). The effect of IPO on GIP may be exaggerated in T2DM patients with impaired insulin sensitivity. Hence, IPO may change the concentrations of gut hormones, postprandial lipaemia, insulinaemic response and CVD related haemostatic markers.

DETAILED DESCRIPTION:
Subjects aged between 30 and 60 years old (male and female) with Type 2 diabetes mellitus (T2DM) will be recruited for this study. A randomized, crossover, double-blind study design will be carried out to investigate the acute effects of high fat meals prepared using palm olein (PO), chemically interesterified palm olein (IPO) and high oleic sunflower oil (HOS) (control) on study subjects with T2DM. Study subjects will have to undergo three postprandial challenges, separated by at least one week interval. Fasting blood sample and duplicate baseline blood samples will be taken in the morning of postprandial day. After that, subjects will be asked to consume a test meal consisting a high fat muffin baked using the aforementioned oils and a milkshake within 10 minutes. After meal, venous blood samples will be taken at time-points 15, 30, 60, 90, 120 min, 3 h, 4 h, 5 h, 6 h and post-heparin plasma 5 min and 15 min for analysis. Pulse wave analysis will be conducted to evaluate central blood pressure and arterial stiffness. Meal appreciation will be assessed by utilising visual analogue scale (VAS) before eating, after eating and at each time-point.

ELIGIBILITY:
Inclusion Criteria:

1. Mild T2DM individuals not planned for medical intervention

   * 7.0 mmol/L ≤ fasting glucose ≤ 11.1 mmol/L
   * 6.5% ≤ HbA1c ≤ 9.0%
   * Not using antihypertensive, lipid lowering, insulin/glucose modulating medication
2. Mild T2DM individuals currently on medical intervention

   * Fasting glucose ≤ 11.1 mmol/L
   * HbA1c ≤ 9.0%
   * Using antihypertensive, lipid lowering or glucose modulating medication
3. Malaysian male or female with T2DM aged between 30 to 60 years old
4. Not using insulin
5. Not having any complications of diabetes
6. No medical history of myocardial infarction, angina, thrombosis, stroke or cancer
7. Haemoglobin levels for females ≥ 11.5 gm/dl and males ≥ 12.5 gm/dl
8. Serum ferritin > 15 µg/l at commencement of study

Exclusion Criteria:

1. Medical history of myocardial infarction, angina, thrombosis, stroke or cancer
2. Underweight (BMI < 18.5 kg/m²)
3. Using insulin
4. Total cholesterol > 7.0 mmol/L
5. Abnormal liver function, renal function and haematology
6. Hypersensitive towards heparin
7. Gastric or lactose intolerance
8. Smoker
9. Pregnancy and lactating
10. Taking alcohol
11. Taking alcohol
12. Haemoglobin levels for females ≤ 11.5 gm/dl and males ≤ 12.5 gm/dl
13. Serum ferritin < 15 µg/l at commencement of study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
6-hour postprandial changes from fasting in glucose-dependent insulinotropic polypeptide (GIP) | 0, 15, 30, 60, 90, 120 min, 3, 4, 5, 6 hour
  To determine the postprandial changes of GIP.

SECONDARY OUTCOMES:
6-hour postprandial changes from fasting in gut hormones | 0, 15, 30, 60, 90, 120 min, 3, 4, 5, 6 h
  To determine the postprandial changes of ghrelin, glucagon-like peptide-1 (GLP-1), peptide YY (PYY) and cholecystokinin (CCK).
6-hour postprandial changes from fasting in insulinaemic response | 0, 15, 30, 60, 90, 120 min, 3, 4, 5, 6 hour
  To determine the postprandial changes of glucose, insulin, C-peptide and non-esterified fatty acid (NEFA)
6-hour postprandial changes from fasting in lipaemia | 0, 1, 2, 3, 4, 5, 6 hour for TAG and apoB48; 6 hour postheparin for LPL; pooled 3, 4, 5 hour for chylomicron and PFA
  To determine the postprandial changes of triacylglycerol (TAG) and apolipoprotein B48 (apoB48).
  To compare lipoprotein lipase (LPL) activity, chylomicron fatty acid composition and plasma fatty acid (PFA) composition across meals.
6-hour postprandial changes from fasting in haemostatic response | 0, 2, 4, 6 hour for FVIIa, PAI-1 and D-dimer; 0, 4 hour for PWA
  To determine the postprandial changes of factor FVII activation (FVIIa), plasminogen activator inhibitor-1 (PAI-1)and D-dimer.
  To compare pulse wave analysis (PWA) across meals.
6-hour changes from fasting hunger rating using visual analogue scale (VAS) | 0, 15, 30, 60, 90, 120 min, 3, 4, 5, 6 hour
  To determine the changes in hunger rating and food satiety

CONTACTS AND LOCATIONS:
Overall Officials: Kim Tiu Teng, PhD, Principal Investigator — Malaysian Palm Oil Board (MPOB)
Locations (5):
- Malaysia (5):
  - Malaysian Palm Oil Board (MPOB), Kajang, Selangor
  - Hulu Langat District Health Office, Kajang, Selangor
  - Sepang District Health Office, Sepang, Selangor
  - Universiti Putra Malaysia, Serdang, Selangor
  - Selangor State Health Office, Shah Alam, Selangor

REFERENCES:
- [Derived] Mo SY, Lai OM, Chew BH, Ismail R, Bakar SA, Jabbar NA, Teng KT. Interesterified palm olein lowers postprandial glucose-dependent insulinotropic polypeptide response in type 2 diabetes. Eur J Nutr. 2019 Aug;58(5):1873-1885. doi: 10.1007/s00394-018-1738-6. Epub 2018 Jun 5. PMID 29872922